CLINICAL TRIAL: NCT06198621
Title: Noninvasive Versus Invasive Methods in Assessment of Hemodynamic Parameters in Respiratory ICU Patients
Brief Title: Hemodynamic Parameters Assessment; Invasive Versus Noninvasive
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Reda, Assistant lecturer in pulmonolgy department, Assiut University
Other Study IDs: cardiometry for hemodynamics
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Output, Low
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: cardiometry — cardiometry is noninvasive method, while swan ganz is invasive method in hemodynamic parameters assessment
  Other Names: pulmonary artery catheter (swan ganz)

SUMMARY:
The study aims at evaluating effectiveness of noninvasive cardiometry in assessment of cardiac parameters in critically ill patients in respiratory ICU in comparison to invasive methods as indirect fick's and thermodilution methods using pulmonary artery catheter.

DETAILED DESCRIPTION:
Patients and methods

A. Study setting The study will be conducted in Assiut University Hospital, in respiratory intensive care unit.

B. Study design This study is a cross-sectional study

C.Methods

Firstly, invasive methods:

The Fick method is a "gold standard" measurement of cardiac output. This method is based on the principle described by Adolfo Fick in 1870, according to which the total uptake or release of a substance by an organ is the product of the blood flow through the organ and the arteriovenous concentration difference of the substance.

The oxygen uptake in the lungs is the product of the blood flow through the lungs and the arteriovenous oxygen content difference. Therefore, the cardiac output, CO, can be calculated using the equation:

CO= VO2/(CaO2-CvO2)

Where VO2 is the oxygen consumption by the lungs and (CaO2-CvO2) is the arteriovenous difference in oxygen. VO2 can be compensated for, based on calculated body surface area (BAS), using equation of = 125 × BSA. The arteriovenous difference is computed by receiving samples of arterial oxygen saturation through arterial blood gases, and mixed venous oxygen saturation through receiving blood from the pulmonary artery using PAC.

Another method is thermodilution, this method uses a special thermistor tipped catheter (Swan-Ganz catheter) inserted from a central vein into the pulmonary artery. A normal saline (temperature 0 degrees Celsius) is injected into the right atrium from a proximal catheter port. This solution causes a decrease in blood temperature, which is measured by a thermistor placed in the pulmonary artery catheter. The pulmonary artery catheter is attached to the cardiac output computer, which displays a curve and calculates output and derived indices automatically.

Secondly, noninvasive methods Electrical cardiometry will be attached to patient using four electrodes. Two electrodes will be on the left side of the neck and the two other electrodes on the left side of the chest opposite to the xiphoid process at the mid-axillary line.

This allow for the continuous measurement of the changes of electrical conductivity within the thorax. By sending low amplitude, high frequency electrical current through the thorax, the resistance that the current faces (due to several factors) is measured. Through advanced filtering techniques, Electrical Cardiometry (EC) is able to isolate the changes in conductivity created by the circulatory system.

This can determine the stroke volume, cardiac output and other hemodynamic indcies.

Another noninvasive method which is used in assessment of cardiac parameters is echocardiography.

D. Action plan and outcomes

1. All patients' data regarding age, gender, sex and essential diagnosis will be taken.
2. Patients' vital signs especially blood pressure and heart rate.
3. Hemoglobin level will be acquired for all patients.
4. Arterial blood gases especially arterial oxygen saturation.
5. Venous blood gases obtained through Swan Ganz catheter.
6. Patients' body surface area using patient height and weight will be obtained
7. All patients will have cardiac parameters assessment using electrical cardiometry.
8. Echocardiography will be recorded for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 18 years old or more.
2. Critically ill patient in respiratory ICU unit with or without hemodynamic instability.

Exclusion Criteria:

1. Presence of active infection at the site of insertion of PCA.
2. Presence of coagulopathy or severe thrombocytopenia.
3. Presence of cardiac arrhythmia or left bundle branch block.
4. Newly inserted pacemaker of the heart.
5. Lack of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Respiratory ICU patients
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of noninvasive cardiometry | 1 year
  To know the effectiveness of noninvasive cardiometry - icon cardiometry - in determining patient's cardiac output and other hemodynamic parameters as stroke volume and cardiac index in comparison to invasive methods using swan ganz catheter as ficks method and thermodilution method. This will be done through computing sensitivity, specificity and accuracy of noninvasive cardiometry.

SECONDARY OUTCOMES:
Abnormal cardiac output in critically ill patients | 1 year
  To know the prevalence of cardiac output abnormalities in critically ill patients in respiratory ICU.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hett DA, Jonas MM. Non-invasive cardiac output monitoring. Intensive Crit Care Nurs. 2004 Apr;20(2):103-8. doi: 10.1016/j.iccn.2004.01.002. PMID 15072778
- [Background] Rodriguez Ziccardi M, Khalid N. Pulmonary Artery Catheterization. 2023 Aug 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482170/ PMID 29489212
- [Background] Evans DC, Doraiswamy VA, Prosciak MP, Silviera M, Seamon MJ, Rodriguez Funes V, Cipolla J, Wang CF, Kavuturu S, Torigian DA, Cook CH, Lindsey DE, Steinberg SM, Stawicki SP. Complications associated with pulmonary artery catheters: a comprehensive clinical review. Scand J Surg. 2009;98(4):199-208. doi: 10.1177/145749690909800402. PMID 20218415
- [Background] Siebenmann C, Rasmussen P, Sorensen H, Zaar M, Hvidtfeldt M, Pichon A, Secher NH, Lundby C. Cardiac output during exercise: a comparison of four methods. Scand J Med Sci Sports. 2015 Feb;25(1):e20-7. doi: 10.1111/sms.12201. Epub 2014 Mar 20. PMID 24646113